CLINICAL TRIAL: NCT07169695
Title: Efficacy and Safety Assessment of T1695 Ophthalmic Suspension, Versus Ciclosporin Ophthalmic Emulsion, in Participants With Moderate to Severe Vernal Keratoconjunctivitis (VKC).
Brief Title: A Study to Compare the Effectiveness and Safety of T1695 Versus Ciclosporin in Participants With Moderate to Severe Vernal Keratoconjunctivitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT1695-201; 2025-521567-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Moderate to Severe Vernal Keratoconjunctivitis
Keywords: Vernal Keratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Slit Lamp Microscopy; Cyclosporine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1695 (Experimental): The participant should instill T1695.
  Interventions: Diagnostic Test: Slit Lamp Examination; Diagnostic Test: Far Best Corrected Visual Acuity (BCVA); Drug: T1695; Diagnostic Test: Corneal fluorescein staining score on modified Oxford scale
- Ciclosporin (Active Comparator): The participant should instill Ciclosporin.
  Interventions: Diagnostic Test: Slit Lamp Examination; Diagnostic Test: Far Best Corrected Visual Acuity (BCVA); Drug: Ciclosporin; Diagnostic Test: Corneal fluorescein staining score on modified Oxford scale

INTERVENTIONS:
Diagnostic Test: Slit Lamp Examination — The participant will have a slit lamp examination
Diagnostic Test: Far Best Corrected Visual Acuity (BCVA) — The participant 's BCVA will be evaluated.
Drug: T1695 — The participant should instill T1695.
  Arms: T1695
Drug: Ciclosporin — The participant should instill Ciclosporin.
  Arms: Ciclosporin
Diagnostic Test: Corneal fluorescein staining score on modified Oxford scale — One drop of fluorescein will be instilled to assess the fluorescein staining score on the modified Oxford scale.

SUMMARY:
The aim of the study is to Compare the Effectiveness and Safety of T1695 Versus Ciclosporin in Participants with Moderate to Severe Vernal Keratoconjunctivitis

ELIGIBILITY:
Main Inclusion Criteria:

* Informed consent signed and dated
* Male or female participant from 4 years to less than 18 years old.
* Participant with grading score of 3 or 4 on the Bonini scale for clinical grading of VKC in each eye.

Main Exclusion Criteria:

Participants must not have any conditions which might exclude them from participating, could interfere with the study, or pose an unacceptable risk to their health.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (Day 1) at Day 29 (Week 4) in Corneal Fluorescein Staining (CFS) grade assessed by the (0-5) modified Oxford scale in the study eye. | From Day 1 to Day 29

IPD SHARING:
Plan to Share IPD: No